CLINICAL TRIAL: NCT07387198
Title: Neoadjuvant Merkel Cell Carcinoma Therapy (Tx) With the PD-1 Inhibitor Cemiplimab - A Randomized, Double-blind, Placebo-controlled, Non-comparative Phase II Study
Brief Title: Neoadjuvant Merkel Cell Carcinoma Therapy (Tx) With the PD-1 Inhibitor Cemiplimab
Acronym: NeoMatryx
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Prof. Gutzmer, Skin Cancer Center Minden, Johannes-Wesling-Klinikum Minden, Germany (Unknown); Prof. Becker, Translational Skin Cancer Research University Duisburg-Essen, Germany (Unknown); Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NeoMatryx
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Merkel Cell Carcinoma, Stage I; Merkel Cell Carcinoma, Stage II; Neoadjuvant Immunotherapy
Keywords: merkel cell carcinoma; sentinel lymph node; PD-1 antibody; skin cancer; Cemiplimab; MCC
MeSH Terms: conditions — Carcinoma, Merkel Cell; Skin Neoplasms | interventions — cemiplimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Cemiplimab) (Experimental): 2 cycles of Cemiplimab (350 mg, i.v., Q3W) followed by sentinel lymph node biopsy
  Interventions: Drug: Cemiplimab 350 mg i.v. on day 1 of every 21 days cycle for 2 cycles
- Arm B (placebo) (Placebo Comparator): 2 cycles of placebo followed by sentinel lymph node biopsy
  Interventions: Drug: Placebo NaCl 0.9% solution i.v. on day 1 of every 21 days cycle for 2 cycles.

INTERVENTIONS:
Drug: Cemiplimab 350 mg i.v. on day 1 of every 21 days cycle for 2 cycles — Patients will receive Cemiplimab 350 mg i.v. on day 1 of every 21 days cycle for 2 cycles
  Other Names: LIBTAYO
  Arms: Arm A (Cemiplimab)
Drug: Placebo NaCl 0.9% solution i.v. on day 1 of every 21 days cycle for 2 cycles. — Patients will receive NaCl 0.9% solution i.v. on day 1 of every 21 days cycle for 2 cycles.
  Arms: Arm B (placebo)

SUMMARY:
The study is a randomized, double blind, placebo-controlled, non-comparative phase II trial that investigates the efficacy of neoadjuvant anti-PD-1 antibody Cemiplimab treatment in patients with clinical stage I or II Merkel cell carcinoma who have have undergone primary tumour excision and are pending sentinel lymph node biopsy.

ELIGIBILITY:
Inclusion criteria

1. Patient has signed informed written consent.
2. Patients is 18 years and older at time of signing of written informed consent
3. Patient has diagnosis of Merkel cell carcinoma in clinical stage II, or in stage I with minimum diameter of 1 cm, with primary tumor already removed and a planned sentinel lymph nodes biopsy still pending.
4. Patient has ECOG performance status 0-2.
5. Patients has adequate laboratory parameters particularly for the blood count, renal and liver function parameters.

   1. Absolute number of neutrophils ≥ 1.5 x 109/L
   2. Platelets ≥ 75 x 109/L
   3. Hemoglobin ≥ 9 g/dL
   4. Total bilirubin ≤ 1.5 times the upper limit of normal (ULN) (patients with Gilbert´s Disease and total bilirubin up to 3x ULN may be eligible after approval from trial's medical expert)
   5. AST (SGOT) and ALT (SGPT) ≤ 3x ULN
   6. AP ≤ 2.5x ULN
   7. Serum creatinine ≤ 2x ULN or creatinine clearance ≥ 40 mL/min
6. Female patients of childbearing potential and male patients with female partners of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 6 months after the last dose of Cemiplimab. Male patients must refrain from donating sperm during this same period. Male patients with a pregnant partner must agree to remain abstinent or to use a condom for the duration of the pregnancy.
7. Patient must be willing to allow translational work-up of tissue samples (PT, sentinel lymph node biopsy).

Exclusion criteria

1. Patient has prior sentinel lymph node removal for the current MCC.
2. Patients received prior treatment with immunotherapy (such as PD-1/PD-L1 or CTL4) or any other systemic anti-tumor (MCC) therapy (incl. investigational therapies)
3. Patient has active or a history of hematological neoplasms including chronic lymphocytic leukemia (CLL), irrespective if these require treatment or not.
4. Patient had prior organ transplantation including allogenic stem-cell transplantation.
5. Patient receives immunosuppressive concomitant medication, EXCEPT for the following:

   i. Intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection).

   ii. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent.

   iii. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
6. Patient has known hypersensitivity to any component of the Cemiplimab formulation as well as a known history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion protein.
7. Patient has active autoimmune or inflammatory disorders.
8. Patient has history of interstitial lung disease.
9. Patient has active infection requiring systemic therapy.
10. Patient has Active infection requiring systemic therapy, including uncontrolled HIV, HBV and HCV infection or diagnosis of immunodeficiency.

    NOTE: Patients are eligible if:
    * Patients have controlled HIV infection with CD4 counts is > 350 cells/μL and viral load is undetectable [HIV RNA PCR]. Patients with controlled HIV infection must be monitored per local standards during the trial.
    * Patients positive for HBV surface antigen have controlled HBV infection receiving anti-viral therapy and with undetectable serum viral load [HBV DNA PCR]. Patients with controlled infection must undergo periodic monitoring of HBV DNA and p must remain on anti-viral therapy for at least 6 months after last dose of Cemiplimab.
    * Patients positive for HCV antibody have controlled HCV infection with undetectable viral load [HCV RNA PCR].
11. Patent received vaccination with any live vaccine (e.g., intranasal flu vaccine) within 4 weeks before the first dose of Cemiplimab or planned vaccination with live vaccine during the trial
12. Female patients, who are pregnant or breast feeding or planning to become pregnant within and 6 months after the end of treatment. Female patients of childbearing potential must have a negative serum β-HCG pregnancy test result within 7 days prior to initiation of study treatment.
13. Patient has evidence of any other disease, neurologic or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of any of the study medications, puts the patient at higher risk for treatment-related complications or may affect the interpretation of study results.
14. Patient has known substance abuse or other psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
15. Patient is legally incapacitated or has limited legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2031-07-31 (Estimated)

PRIMARY OUTCOMES:
Nodal micrometastases-free rate | up to 36 months
  rate of patients without nodal micrometastases after 2 cycles of treatment, determined by sentinel lymph node biopsy

SECONDARY OUTCOMES:
Recurrence-free survival | up to 66 months
  time from randomization until date of the first of the following events: MCC progression, MCC recurrence, and MCC-related death
Overall survival | up to 66 months
  time from randomization until date of death from any cause
Disease specific survival | up to 66 months
  time from randomization until date of MCC-related death
Quality of life using FCRI-SF questionnaire | up to 66 months
  Quality of life determined using the FCRI-SF questionnaire
Safety (AEs and SAEs) | up to 66 months
  incidence, nature, causality, frequency, timing and severity of adverse events using NCI CTCAE 5
Quality of life using the mFACT-M questionnaire | up to 66 months
  Quality of life determined using the mFACT-M questionnaire

OTHER OUTCOMES:
Investigation of prognostic and predictive biomarkers to estimate the risk of lymph node metastases and signs of immune activation in the sentinel lymph nodes | up to 66 months
  Biosamples will be used to determine the correlation of identified biomarkers with clinical outcome, i.e., nodal metastases-free rate, RFS, OS

CONTACTS AND LOCATIONS:
Overall Officials: Salah Al-Batran, Prof. Dr., Study Director — Institut für Klinische Krebsforschung IKF GmbH; Ralf Gutzmer, Prof. Dr. med., Principal Investigator — Johannes Wesling Klinikum Minden; Juergen C. Becker, Prof. Dr. Dr., Principal Investigator — Translational Skin Cancer Research University Duisburg-Essen, Germany
Locations (14):
- Germany (14):
  - Nationales Centrum für Tumorerkrankungen, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Mannheim, Mannheim, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Regensburg, Regensburg, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg, Hamburg
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Klinikum Bielefeld, Bielefeld, North Rhine-Westphalia
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Johannes Wesling Klinikum Minden, Minden, North Rhine-Westphalia
  - Universitätsmedizin Mainz, Mainz, Rhineland-Palatinate
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Helios Klinikum Erfurt, Erfurt, Thuringia

IPD SHARING:
Plan to Share IPD: No